CLINICAL TRIAL: NCT04828252
Title: The Effects of Low Level Laser Intervention on Muscular Strength for Individuals With Knee Osteoarthritis
Brief Title: Low Level Laser Intervention for Individuals With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A-ER-109-187
Record Dates: First submitted 2021-02-03; First posted 2021-04-02 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-02

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 808nm (Experimental): The wavelength of this experimental group was 808nm, total power: 3.6W, 15 minutes a session, 3 times a week for 8 weeks
  Interventions: Device: Low level laser treatment
- 660nm (Active Comparator): The wavelength of this experimental group was 660nm, total power: 3.6W, 15 minutes a session, 3 times a week for 8 weeks
  Interventions: Device: Low level laser treatment
- Control (Placebo Comparator): The wavelength of control group, total power: 0.0072W, 15 minutes a session, 3 times a week for 8 weeks
  Interventions: Device: Low level laser treatment

INTERVENTIONS:
Device: Low level laser treatment — The intervention protocol includes 2 wavelength as the experimental group, each of the were 808nm, 660nm, and 1 placebo intervention which output total power is only 0.0072W.

SUMMARY:
The purpose of this study was to investigate the intervention effects of low level laser for knee OA group

ELIGIBILITY:
Inclusion Criteria:

* The severity of osteoarthritis was defined by the Kellgren-Lawrence system as grade 2 - grade 3

Exclusion Criteria:

* Uncontrolled hypertension
* Malignant tumor
* Skin cancer
* Pregnant
* Dysesthesia
* Pacemaker inplement
* Cognitive problem
* Fall record within 6 months
* Dysfunction of blood coagulation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2021-06-04 (Actual)

PRIMARY OUTCOMES:
Changes of muscular strength of thigh measured by handheld dynamometer | Baseline and after treatment, 8 weeks intervention
  Muscular strength of the knee extensor and flexor on both sides and will be normalized by the body weight of participants' (lb/kg)

SECONDARY OUTCOMES:
Changes of walking speed measured by the stop watch | Baseline and after treatment, 8 weeks intervention
  40-m walk test, participants are instructed to walk as fast as they could, investigator records the time they spend. (seconds)
Changes of stair climbing ability measured by the stop watch | Baseline and after treatment, 8 weeks intervention
  stair climbing test, participants are instructed to climb stairs with a total height of 180 cm as fast as they could, investigator records the time they spend. (seconds)
Changes of chair stand ability, the stop watch will be used to measure time and investigators count the time that participants complete | Baseline and after treatment, 8 weeks intervention
  sit-to-stand test, participants are instructed to repeat chair stand movement as fast as they could, investigator records the times they complete. (times)
Changes of dynamic balance ability measured by the stop watch | Baseline and after treatment, 8 weeks intervention
  timed UP&Go test, participants are instructed to stand up from a chair and walk as fast as they could for 3 meters and back to the chair, investigator records the time they spend. (seconds)

OTHER OUTCOMES:
Changes of joint range of motion measured by the goniometer | Baseline and after treatment, 8 weeks intervention
  Joint range of motion of the hip flexion, internal and external rotation, knee flexion, extension on both sides(degrees)

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Feng Lin, Ph.D, Study Chair — Department of Physical Therapy, National Cheng-Kung University
Locations (1):
- Department of Physical Therapy, National Cheng-Kung University, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided